CLINICAL TRIAL: NCT04613713
Title: Effectiveness and Cost-utility of Somatocognitive Therapy Versus Treatment as Usual for Provoked (Localized) Vestibulodynia - a Randomized Clinical Trial (ProLoVe Study)
Brief Title: Somatocognitive Therapy in Treatment of Provoked (Localized) Vestibulodynia - Randomized Clinical Trial (ProLoVe Study)
Acronym: ProLoVe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29295
Record Dates: First submitted 2020-10-26; First posted 2020-11-03 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-04

CONDITIONS: Vulvodynia; Vestibulodynia
Keywords: Provoked vestibulodynia; Dyspareunia; Somatocognitive therapy; Physiotherapy; Randomised clinical trial; Women's health; Sexual dysfunction; Pain management
MeSH Terms: conditions — Vulvodynia; Dyspareunia; Sexual Dysfunction, Physiological; Agnosia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Parallel group randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: Statistician analyzing the data will be blinded for group belonging
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Somatocognitive physiotherapy (Experimental): Somatocognitive therapy is a multi-modal physiotherapy intervention utilized for women with longstanding chronic pelvic pain and provoked vestibulodynia developed at the beginning of the 2000s as a collaboration between the department of psychosomatic medicine, Oslo University Hospital (OUH) and department of physiotherapy (OsloMet)
  Interventions: Other: Somatocognitive physiotherapy
- Treatment as usual (Active Comparator): The participants randomized to the treatment as usual group will follow available treatment options based on the current recommendations from Vulva clinic at Oslo University Hospital, a center that is specialized in treatment of vulvar conditions.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Other: Somatocognitive physiotherapy — The main intervention areas include:
  1. education about the PVD, healthy vulvo-vaginal and sexual behaviors, nature of chronic pain and factors influencing pain intensity
  2. bodily exercises and techniques increasing body awareness, ability to relax and control muscle tension and respiration pattern in different situations
  3. techniques to cope with emotions and thoughts related to bodily experiences and to PVD
  4. structured homework assignments promoting application of the learned techniques in daily situations and gradual exposure of the patient to activities associated with pain.
  Participants will be offered maximally 15 treatment sessions. No minimal number of sessions is set. Treatment will be conducted by female physiotherapists experienced in treating long-standing pain conditions.
  Arms: Somatocognitive physiotherapy
Other: Treatment as usual — The participants will follow the current treatment advice as recommended by the Vulva Clinic at OUH, a tertiary health care center specialized in treatment of vulvar disorders. Advice include guidance about the management of PVD as a condition, use of medication, physiotherapy, sexologist and psychological counseling, usage of internet resources (vulva.no) and others. Participants will be free to pursue treatment options of their choice. The type of treatment, number of treatments and medication usage will be monitored by bi-weekly electronic forms during the whole study period.
  Arms: Treatment as usual

SUMMARY:
This is a two-arm randomized clinical trial assessing effectiveness of somatocognitive therapy versus treatment as usual for provoked vestibulodynia (PVD). PVD is a common, but under-treated persistent pain condition, mostly affecting young women in their late teens and early 20s. It is the most frequent cause of pain during sexual intercourse affecting around 10% of women in the general population. There are no generally accepted evidence-based guidelines for the medical management of PVD. The most commonly used treatments are topical (85%), physiotherapy (52%), and oral medications (45%). High quality randomized clinical trials testing effectiveness of various therapy approaches are urgently needed.

Somatocognitive therapy SCT is a multi-modal physiotherapy approach developed for alleviating musculoskeletal persistent pain conditions. SCT has been previously evaluated in the treatment of women with chronic pelvic pain.

In the current study, 128 women with PVD will be randomized into SCT and treatment as usual (TAU) group. Participants will be assessed at baseline, after 6 months and after 12 months. The main outcome will be changes in female sexual function index scored at 12 months follow up. Secondary outcomes include pain intensity as assessed by a tampon test as well as a number of questionnaires recording different aspects of emotional and cognitive functioning. In addition cost-effectiveness analysis of SCT versus TAU will be performed.

Participants in the SCT group will receive up to 15 therapy sessions and will additionally be offered one booster session at 6 months after treatment ending. TAU group will follow treatment options of their own choice based on recommendations from the Vulva clinic at Oslo University Hospital, a center that is specialized in treating women with vulvar pain conditions.

DETAILED DESCRIPTION:
Objectives:

The main objectives of the ProLoVe study are:

1. To assess clinical effectiveness of somatocognitive therapy (SCT) versus treatment as usual (TAU) in provoked vestibulodynia (PVD).
2. To identify prognostic factors associated with treatment outcome
3. To assess cost-effectiveness and cost-utility of SCT vs TAU.

Study design:

The study is a two-arm, single center randomized clinical trial with a 1:1 allocation ratio, recruiting patients with PVD diagnosis. The participants will be randomized to either somatocognitive therapy (SCT) or treatment as usual (TAU) group after baseline assessment. Randomization will be stratified by type of PVD (primary or secondary), since primary PVD is considered to be more treatment resistant.

Recruitment procedure:

Participants' eligibility will be evaluated by the medical specialist in gynecology or dermatology. During medical consultation an eligible patient will be verbally informed about the study and receive an information leaflet about the project. Number of eligible patients informed about the study, will be registered. Interested women will contact the primary investigator who will set up a meeting. Detailed information about the trial, the assessment instruments and existing treatment options will be provided. Women willing to pursue study participation will sign an informed consent.

Randomization and blinding:

An administrative coordinator, not directly involved in the study, will be responsible for randomization of the participants using a computer random number generator, and will be responsible for the secure storage of randomization results. The participants will be randomized to either somatocognitive physiotherapy (SCT) or treatment as usual group (TAU) at 1:1 allocation rate. Randomization will be stratified by severity (primary/secondary PVD). Blinding of the participants regarding group belonging is not possible.

Data collection:

All quantitative instruments will be distributed as electronic forms (nettskjema.no) and directly transferred to the Service for Sensitive Data (TSD). Choice and implementation of assessment instruments is based on the Recommendations for the study of the vulvar pain in women, part I: review of assessment tools (Rosen et al. 2020), feedback from participants from the feasibility study and discussions with user representative (former PVD patient). Three assessment time points are planned: baseline, 6 months follow up, and 12 months follow up.

Sample size assessment:

Power analysis suggests that 128 participants split equally between two study arms will be enough to reveal the between group difference in total FSFI score changes, from baseline to 12 months follow-up, of at least 3 points (SD = 6.0) as statistically significant, using α = 0.05 and 1-β = 0.8. In a feasibility study (n=10) an average of 6 points improvement on FSFI in course of 8 months in patients treated with SCT was observed.

Data analysis:

Objective 1: To assess clinical effectiveness of somatocognitive therapy (SCT) versus treatment as usual (TAU) in provoked vestibulodynia (PVD).

Hypothesis 1: In treatment of PVD, the effectiveness of somatocognitive therapy is not significantly different from treatment as usual as evaluated by changes in FSFI total score from baseline to 12 months follow-up

Independently, a senior statistician and PhD student blinded to treatment group will perform intention to treat analyses of the treatment effect on the primary outcome by using linear mixed model for repeated measures.

Subgroup analysis (objective 1) Some of the women with PVD do not engage in penetrative sex and thus score 0 at the FSFI pain sub-scale. This influences the psychometric properties of FSFI and it is recommended to exclude the pain sub-scale from the analysis in those cases. Therefore, additional analyzes will be performed on the subgroups of women who did and did not have penetrative sex during the 4 weeks prior to FSFI completion using the same statistical approaches as for hypothesis 1.

Objective 2: To identify prognostic factors associated with treatment outcome

For prognostic analyses, changes in FSFI scores between baseline and 12 months follow up as the dependent variable will be used. Further, an association model to assess possible associations between selected variables and the main outcome will be constructed. The variables that reached the level of significance of at least 0.10 in univariate analyses will be entered into multiple regression models. To avoid over-fitting, at most, one variable per 10 events will be included. In addition, highly correlated covariates (>0.7) will not be included in the final model.

Objective 3: To assess cost-effectiveness and cost-utility of SCT vs TAU.

The cost-effectiveness analysis will be carried out from a healthcare and society perspective, comparing the treatment effect and health utilities by using the EuroQoL 5D (EQ-5D-5L) utility index. Health gains will be expressed as quality-adjusted life years (QALYs) derived from the EQ-5D-5L utility scores. Costs to the healthcare system and society (production loss) due to PVD will be estimated based on data recorded at the follow-ups including visits to general practitioner, medical specialist, physical therapist, manual therapist or other physical therapy specialist, and other therapists (e.g. chiropractor, osteopath, psychologist); number of days of hospitalization and/or rehabilitation; use of medication). Data concerning production loss will include work status in terms of working time (percentage of position), partial sick leave (percentage, duration, and reason), complete sick leave (duration and reason), disability pension (percentage, duration, and reason), unemployment (yes, no), and student/other/unknown (yes, no).

Secondary analysis

Proportion comparisons of women who experienced successful treatment outcome in SCT and TAU group will be analyzed using global perceived effect scale at 12 months follow up applying logistic regression for repeated measures. Within and between group differences in other secondary outcomes will be evaluated using linear mixed model for repeated measures.

Exploratory analysis in TAU group Participants in the TAU group may choose a variety of different treatment options, e.g. other types of physiotherapy, osteopathy, chiropractor treatment, etc. Exploratory analysis will be conducted to identify the most promising treatments with respect to improvement on the FSFI using repeated measures analysis of variance. The goal of these analyses is to identify candidate treatments for future studies.

In all analyses, the between-group mean differences with 95% confidence intervals (CI) or odds ratio (OR) with 95% CI for categorical outcomes will be reported. Missing data will be replaced using multiple imputation methods.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of provoked vestibulodynia
* Age: 18 to 35
* Must understand Norwegian well enough to be able to complete questionnaires
* Must be able to attend treatment in Oslo, Norway

Exclusion Criteria:

* Active infection in the vulvar region
* Dermatologic lesion in the vulvar region
* Presence of diagnostically confirmed psychiatric condition that necessitate treatment by a medical specialist in psychiatry of clinical psychology

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 128 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in female sexual function index (FSFI) (Rosen et al. 2000) | Baseline, 6 and 12 months follow up
  A multidimensional scale assessing key dimensions of female sexual function. The FSFI is a 19-item self-report questionnaire designed to measure sexual functioning in women. It assesses six domains of sexual function: sexual desire, sexual arousal, lubrication, orgasm, satisfaction, and pain (i.e., pain associated with vaginal penetration). Higher scores indicate better sexual functioning.

SECONDARY OUTCOMES:
Change in Participant Perceived Improvement (PGIC) (Dworkin et al. 2005) | 6 and 12 months follow up
  Participants are asked to rate on a 7-points Likert scale how much their condition has changed since baseline measurement. Answering alternatives: very much improved, much improved, minimally improved, no change, minimally worse, much worse, very much worse
Change in the tampon test (Foster et al. 2009) | Baseline, 6 and 12 months follow up
  The tampon test measures vulvar pain intensity during insertion and removal of a standard sanitary tampon. At each assessment time (baseline, 6 and 12 months follow up), the test will be performed three times at home during a 7-day period, on days 1, 4 and 7. A mean value of these 3 measurements will be used as a measure of pain sensitivity. Pain intensity is recorded on the Numeric Rating Scale (0-10) where 0 is no pain and 10 is the worst pain imaginable.
Change in recalled pain intensity during intercourse | Baseline, 6 and 12 months follow up
  Participant is asked to score on a Numeric Rating Scale (0-10) how intense was the pain during last intercourse, where 0 is no pain and 10 is the worst pain imaginable.
Change in Vulvar Pain Assessment Questionnaire (VPAQ) (Dargie et al. 2017) - life interference | Baseline, 6 and 12 months follow up
  VPAQ is developed to assist in the assessment and diagnosis of vulvodynia. Life interference sub-scale describes impact of vulvodynia on daily living. It consists of 11 questions addressing different domains of daily functioning. Each question is scored on a 6-points Likert scale with a higher score indicating higher negative impact of vulvodynia on daily activities
Change in Vulvar Pain Assessment Questionnaire (VPAQ) (Dargie et al. 2017) - coping strategies | Baseline, 6 and 12 months follow up
  VPAQ - coping strategies sub-scale consists of 12 statements describing different pain-coping strategies. Each statement is scored on a 5-points Likert scale referring to how often a specific strategy is used. A higher score indicate more frequent use of a given strategy.
Change in vulvodynia related self-efficacy | Baseline, 6 and 12 months follow up
  The scale will be assessed to record participant's belief in her ability to cope with the vulvodynia symptoms on her own. The scale is based on one question scored on 5-points Likert scale with higher scores indicating higher belief in woman's ability to cope with her symptoms.
Change in pain catastrophizing scale (Fernandes et al. 2012) | Baseline, 6 and 12 months follow up
  The pain catastrophizing scale is a self-report measure consisting of 13 items scored from 0 to 4. The higher the score, the more catastrophizing thoughts are present. It assesses an impact of negative cognition's and catastrophizing on pain experience. This version of the scale has been specifically adapted for pain related to vulvodynia.
Change in Rumination Response Scale (RRS-10) (Parola et al. 2017) | Baseline, 6 and 12 months follow up
  Rumination and worry express a method of coping with negative emotions and feelings that is characterized by self-focused attention, repetitive focus on negative emotions and self-reflection. RSS-10 includes 10 questions scored on a 4-points Likert scale. The higher scores indicate more worry and rumination.
Change in Hopkins Symptoms Check List (HSCL-25) (Derogatis et al.1974) | Baseline, 6 and 12 months follow up
  HSCL-25 evaluates psychological distress related to the anxiety and depression symptoms. It consists of 25 questions scored on a 4-points Likert scale. Higher scores indicate higher levels of psychological distress.
Change in EQ-5D-5L (Herdman et al. 2011) | Baseline, 6 and 12 months follow up
  EQ-5D-5L is used to assess health related quality of life and/or cost-effectiveness of assessed interventions. It consists of 5 domains scored on 5-points Likert scale with higher scores indicating lower quality of life. Additionally 100 points NRS scale is used for evaluation of current health status with higher score indicating better health.

CONTACTS AND LOCATIONS:
Overall Officials: Slawomir Wojniusz, Phd, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan University, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Foster DC, Beth Kotok M, Huang LS, Watts A, Oakes D, Howard FM, Stodgell CJ, Dworkin RH. The tampon test for vulvodynia treatment outcomes research: reliability, construct validity, and responsiveness. Obstet Gynecol. 2009 Apr;113(4):825-832. doi: 10.1097/AOG.0b013e31819bda7c. PMID 19305326
- [Background] Dargie E, Holden RR, Pukall CF. The Vulvar Pain Assessment Questionnaire: Factor Structure, Preliminary Norms, Internal Consistency, and Test-Retest Reliability. J Sex Med. 2017 Dec;14(12):1585-1596. doi: 10.1016/j.jsxm.2017.10.072. PMID 29198513
- [Background] Fernandes L, Storheim K, Lochting I, Grotle M. Cross-cultural adaptation and validation of the Norwegian pain catastrophizing scale in patients with low back pain. BMC Musculoskelet Disord. 2012 Jun 22;13:111. doi: 10.1186/1471-2474-13-111. PMID 22726668
- [Background] Parola N, Zendjidjian XY, Alessandrini M, Baumstarck K, Loundou A, Fond G, Berna F, Lancon C, Auquier P, Boyer L. Psychometric properties of the Ruminative Response Scale-short form in a clinical sample of patients with major depressive disorder. Patient Prefer Adherence. 2017 May 12;11:929-937. doi: 10.2147/PPA.S125730. eCollection 2017. PMID 28553085
- [Background] Derogatis LR, Lipman RS, Rickels K, Uhlenhuth EH, Covi L. The Hopkins Symptom Checklist (HSCL): a self-report symptom inventory. Behav Sci. 1974 Jan;19(1):1-15. doi: 10.1002/bs.3830190102. No abstract available. PMID 4808738
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Rosen NO, Bergeron S, Pukall CF. Recommendations for the Study of Vulvar Pain in Women, Part 1: Review of Assessment Tools. J Sex Med. 2020 Feb;17(2):180-194. doi: 10.1016/j.jsxm.2019.10.023. Epub 2019 Dec 4. PMID 31812684